CLINICAL TRIAL: NCT02807168
Title: NT-proBNP in the Management of Discharged Patients With Acutely Decompensated Heart Failure and Preserved Ejection Fraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Collaborators: Juan Cinca Cuscullola (Unknown); Pablo García Pavía (Unknown); Manuel Martinez Selles (Unknown); Antoni Bayés Genís (Unknown); Alfonso Varela Román (Unknown); Pedro Luis Sánchez Fernández (Unknown)
Responsible Party: Principal Investigator, Domingo A. Pascual Figal, University Professor, MD, PhD, Hospital Universitario Virgen de la Arrixaca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NICE-preserve
Record Dates: First submitted 2016-06-03; First posted 2016-06-21 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Heart Failure; Preserved Left Ventricular Ejection Fraction
MeSH Terms: conditions — Heart Failure | interventions — pro-brain natriuretic peptide (1-76)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Control Group
- Usual care plus NT-proBNP (Experimental): Experimental Group
  Interventions: Other: NT-proBNP (Cardiac Biomarkers)

INTERVENTIONS:
Other: NT-proBNP (Cardiac Biomarkers)
  Arms: Usual care plus NT-proBNP

SUMMARY:
Acute decompensated heart failure (ADHF) is a health problem of great magnitude, because it is the most frequent cause of hospitalization of patients over 65 years old. Of these patients, more than 50% will be readmitted within the next six months with the consequent worsening prognosis, increased mortality and high costs associated. In fact, two-third parts of the costs of this condition are due to hospitalizations. Hence the increased importance of ADHF and its associated hospitalizations as an essential event in the natural history of the disease on to address therapeutic efforts.

However, at the present time there is a change of scenario that makes that more than half of these patients show HF with preserved ejection fraction (PEF), so that acute heart failure with preserved ejection fraction (AHF-PEF) is a fact with high prevalence and epidemiological relevance. To this the investigators must add that, unlike patients with depressed EF, HF-PEF has no therapeutic strategies that may have proven a recovery of the affected patients. All this makes that overall heart failure with PEF and AHF-PEF represent a major health problem.

However, despite of the lack of effective treatments, there are also opportunities for improvement both in terms of morbidity and mortality that should be evaluated. Rather than looking for therapies or new specific drugs, these opportunities may be in the use of management strategies among which the use of biomarkers and their monitoring could be key. In this regard, NT-proBNP has been shown to correlate with severity and prognosis, including the risk of decompensation. Nevertheless, whilst the latest guidelines for heart failure management recommend its use in the diagnosis of HF, the use of biomarkers to monitor and guide treatment has not been included yet.

The assumption of this study is that the use of NT-proBNP may serve as a therapeutic and management guideline for the in-patient with HF-PEF who is to be discharged, allowing a reduction of decompensations and hospitalizations as well as a better functional situation at 6 months.

Several criteria have been proposed to define the syndrome of HFpEF according to the 2013 ACCF/AHA Heart Failure Guideline including (a) clinical signs or symptoms of HF; (b) evidence of preserved or normal LVEF; and (c) evidence of abnormal LV diastolic dysfunction that can be determined by Doppler echocardiography or cardiac catheterization The assay N-terminal proB-type natriuretic peptid is indicated as an aid in the diagnosis of individuals suspected of having congestive heart failure and detection of mild forms of cardiac dysfunction. The test also aids in the assessment of heart failure severity in patients diagnosed with congestive heart failure. This assay is further indicated for the risk stratification of patients with acute coronary syndrome and congestive heart failure, and it can also be used for monitoring the treatment in patients with left ventricular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are discharged after hospitalizations for AHF which is defined by:

   * Dyspnea at rest or with minimal effort
   * Pulmonary congestion on chest X ray
   * NT-pro-BNP levels in the first 24 hours after admission:

   <50 years: >450 pg/ml 50-75 years: >900 pg/mL >75 years: >1800 pg/mL
2. -Administration of at least 40 mg IV furosemide (or equivalent) at admission
3. -Preserved ejection fraction (LVEF>50%) in echocardiography performed at admission and evidence of diastolic dysfunction defined according to following parameters

   * e´ <8 cm/s septal or <10 cm/s lateral (TDI mitral annulus)
   * E/e' ratio >15
   * A mitral-A pulmon > 30 msg
   * Left atrial volumen index≥34 mL/m2
   * left ventricular mass index >95 g/m2 (woman) o >115 g/m2 (man)
4. -Ability to sign the informed consent

Exclusion Criteria:

1. Significant lung disease demonstrated by spirometry
2. Life´s prognosis < 6 months
3. Patients who does not have adhesion at the different visits of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2015-06; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Decrease of rehospitalizations due to acute heart failure at 6 months after discharge. | 6 months
  To assess if a clinical management strategy that includes the monitoring of NT-proBNP concentrations after hospital discharge of patients with AHF-PEF reduces rehospitalizations due to AHF at 6 months after discharge (defined as unplanned hospital admission lasting for at least 24 h and due to HF decompensation).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Virgen de La Arrixaca, Murcia, Spain